CLINICAL TRIAL: NCT03163212
Title: Safety and Tolerability of Lactoferrin/FOS in Very Low Birth Weight Infants
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Virginia (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, David A Kaufman, Neonatologist, University of Virginia
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19804
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Safety Issues; Tolerance; Very Low Birth Weight Infant
Keywords: Lactoferrin/FOS Supplementation

STUDY DESIGN:
Intervention Model Description: Dose escalation design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lactoferrin/FOS 100mg/kg (Experimental): 100 mg/kg enteral administration daily for 30 days
  Interventions: Dietary Supplement: Lactoferrin/FOS
- Lactoferrin/FOS 200mg/kg (Experimental): 200 mg/kg enteral administration daily for 30 days
  Interventions: Dietary Supplement: Lactoferrin/FOS
- Lactoferrin/FOS 300mg/kg (Experimental): 300 mg/kg enteral administration daily for 30 days
  Interventions: Dietary Supplement: Lactoferrin/FOS

INTERVENTIONS:
Dietary Supplement: Lactoferrin/FOS — Bovine Lactoferrin/FOS 100mg/ml dissolved in sterile water
  Other Names: BF100

SUMMARY:
This study will examine the safety and tolerability of supplementation with bovine lactoferrin with fructo-oligosaccharide a simple sugar in very low birth weight infants. Lactoferrin is a major whey protein in mother's milk and plays a role in promoting a mature and healthy gut. It also has antimicrobial and immunomodulation activities.

DETAILED DESCRIPTION:
Aim 1: To evaluate the safety and tolerability of three different lactoferrin/FOS doses in preterm infants

1. Lactoferrin/FOS related adverse events and serious adverse events
2. Time reaching full feeds while receiving lactoferrin/FOS (120 ml/kg/day)
3. Episodes of not receiving enteral feedings for > 24 hours once feeding is initiated

Aim 2: To evaluate lactoferrin/FOS absorption and excretion

1. Examine lactoferrin/FOS levels in saliva, urine, plasma, and stool
2. Examine lactoferrin levels in materal and human donor milk

Aim 3: To evaluate the effect of lactoferrin/FOS on the intestinal microbiome structure

ELIGIBILITY:
Inclusion Criteria:

* < 15 days of age and receiving enteral feedings
* < 1500 grams birth weight
* < 37 weeks gestation

Exclusion Criteria:

* Congenital bowel obstruction (esophageal, duodenal, small bowel or anal atresias, Hirschsprung disease, malrotation)
* Known necrotizing enterocolitis or bowel perforation

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Definitely related study solution serious adverse event | 30 days while receiving study solution

SECONDARY OUTCOMES:
Day after birth to reach 120ml/kg of enteral feeds | 30 days while receiving study solution
Number of days not receiving any feedings after lactoferrin/FOS administration | 30 days while receiving study solution

IPD SHARING:
Plan to Share IPD: Undecided
Specimens which have been unidentified may be shared with outside labs for analysis